CLINICAL TRIAL: NCT06042933
Title: Early Oral Feeding Versus Traditional Delayed Oral Feeding Post-perforated Peptic Ulcer Repair: A Comparative Study in Egyptian Tertiary Health Care Center
Brief Title: Early Oral Feeding Versus Traditional Delayed Oral Feeding Post-perforated Peptic Ulcer Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Elshwadfy Nageeb, lecturer of general surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-96-2023
Record Dates: First submitted 2023-07-28; First posted 2023-09-21 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Peptic Ulcer Perforation
MeSH Terms: conditions — Peptic Ulcer Perforation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): early oral intake 6 hours postoperative.
  Interventions: Other: Post operative early oral feeding
- Group B (Active Comparator): delayed oral intake after 72 hours
  Interventions: Other: Traditional delayed oral Feeding Post-perforated Peptic Ulcer Repairs

INTERVENTIONS:
Other: Post operative early oral feeding — To start oral feeding 6 hours after perforated peptic ulcer repairs
  Arms: Group A
Other: Traditional delayed oral Feeding Post-perforated Peptic Ulcer Repairs — To start oral feeding after 48 hours
  Arms: Group B

SUMMARY:
This study aims to evaluate safety and benefits of early oral feeding compared to traditional delayed oral feeding in patients undergoing perforated peptic ulcer repairs. Study population & Sample size :(

DETAILED DESCRIPTION:
Study Design:

This study is a single-center, prospective, parallel arm, randomized controlled trial. Patients will be randomly assigned in 1:1 ratio to receive either delayed oral feeding or early oral feeding.

Methods:

Patients will be randomly assigned into two groups. Group A patients followed an early oral feeding protocol(12 hours), and Group B received delayed oral feeding (72 hours).

Outcome parameter :

The outcomes are incidence of postoperative complications including Postoperative repair leakage, Infection-related postoperative complications , Number of days of hospital stay and return of bowel function and Diet intolerance.

ELIGIBILITY:
Inclusion Criteria:

- All consecutive patients, of age 18 years and above, who were

presented to the emergency surgical team and were diagnosed with perforated duodenal ulcer by surgicalteam, were recruited and assessed for eligibility.

Exclusion Criteria:

* • Preoperative refractory septic shock on admission.

  * Delayed presentation more than 24 hours.
  * The presence of neuropsychiatric disease, pregnant and lactating women.
  * Predisposing factors for impaired wound healing (e.g., currently using immunosuppressive agents, or chronic use of steroids), the presence of HIV.
  * American society of anesthesiologists grade iii/iv, or had an alternative perioperative diagnosis.
  * Intraoperatively, after randomization, patients were excluded based on the following criteria: perforated duodenal ulcer ≥20 mm, consistent with malignant ulcers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
number of days of hospital stay | Up to 10 days
  number of days of hospital stay
days needed for frist Bowel motion | 7 days
  number of days before frist bowel motion

SECONDARY OUTCOMES:
incidence of Post operative repair leak | 30 days
  number of Post operative repair leaks
severity of operative pain measured by Visual Analogue Scale (VAS) | 7 days
  from 1 to 10 1 indicated minimum pain and 10 maximum pain
INCIDENCE OF postoperative nausea and vomiting (PONAV) | 7 days
  number of cases with postoperative nausea and vomiting (PONAV)
incidence of Surgical site infection | 30 days
  number of cases complicated with surgical site infection
incidence of Pulmonary complications | 30 days
  number of cases complicated Pulmonary complications
incidence of Ryle reinsertion | 7 days
  number of cases complicated Ryle reinsertion
number of Readmission cases | 30 days
  number of cases complicated Readmission cases

CONTACTS AND LOCATIONS:
Overall Officials: mohammed elshwadfy, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt